CLINICAL TRIAL: NCT04830605
Title: Feasibility Test of the Treatment Program iACT-by Proxy - a Single Case Experimental Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Katrine Ingeman Beck, Psychologist, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-296-20
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Anxiety State; Anxiety Disorders
Keywords: Internet-based treatment; Single-case experimental design
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a single-case experimental design with multiple baselines. This means the participants have different baseline lengths but the same intervention and follow-up period and that they all receive the same intervention. The baseline and intervention period serves as two study conditions, a control (baseline) and a treatment condition (intervention) with N equally spaced measurement occasions. The baseline length is randomly assigned to the participants and serves as each participants' own control-condition. This makes it possible to have a small number of participants. If the intervention shows effect a change in the anxiety level will be detected during the intervention period regardless of when the intervention-period was initiated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Internet-delivered treatment for parents with health anxiety on behalf of their child. Eight weeks with therapist support.
  Interventions: Behavioral: Internet-based treatment

INTERVENTIONS:
Behavioral: Internet-based treatment — The intervention is an internet-based psychotherapy treatment with eight modules based on acceptance and commitment therapy and with written therapist contact through eight weeks.

SUMMARY:
Health anxiety by proxy is defined as parents' obsessive worries about their child's health. It is a newly described phenomenon, where the parent has persistent and distressing fears that his or her child may suffer from a serious disease that is being overlooked. These intrusive thoughts may lead to excessive attention directed towards their child's body and a tendency to interpret natural bodily sensations as unnatural and abnormal. As a consequence, parents with health anxiety by proxy may repetitively perform bodily inspections of their child. Besides the stress related to worrying about your child's health, the condition can also cause frequent and unnecessary medical examinations of the child. As a possible consequence of this parental behavior, the child may be at risk of developing similar maladaptive illness behaviors, illness perceptions and illness worries. Currently, the phenomenon is widely overlooked and no treatment for health anxiety by proxy exists.

The aim of the study is to test the feasibility and possible effect of an internet-based treatment program for health anxiety by proxy (iACT-by-proxy) using a single-case experimental design.

Design The iACT-by-proxy is being tested in a single-case experimental design with multiple baselines. In a multiple baseline design the participants have different baseline lengths but the same intervention and follow-up period. The rationale behind the different baseline lengths is that it will be evident if target outcome measures change at intervention entry, but not during baseline. Thus the participants' baseline-period functions as their own control.

Hypotheses

* Patients will report a significant decrease in selected self-report measures of health anxiety by proxy answered every other day when comparing the baseline period to the interven-tion period.
* Patient self-report measures of health anxiety by proxy, emotional distress, and illness perception and catastrophizing when the child has symptoms will have decreased after intervention.

Participants Parents assessed with health anxiety by proxy with children under 18years.

Recruitment Participants are assessed with health anxiety by proxy using the Health Anxiety by Proxy Scale (HAPYS).Participants self-refer to the project through the webpage www.helbredsangst.dk. After diagnostic video-interview they are included in the project.

DETAILED DESCRIPTION:
Background

Health anxiety by proxy is a newly described phenomenon, where the parent has persistent and distressing fears that his or her child may suffer from a serious disease that is being overlooked. These intrusive thoughts may lead to excessive attention directed towards their child's body and a tendency to interpret natural bodily sensations as abnormal. As a consequence, parents with health anxiety by proxy may repetitively perform bodily inspections of their child or have medicial examinations conducted (1, 2). As a possible consequence of this parental behavior, the child may be at risk of developing similar maladaptive illness behaviors, illness perceptions and illness worries(3).

Research on parents suffering from health anxiety has found evidence of health anxiety symptoms being transmitted from parent to child (4, 5) indicating that the parent's response to the child's health complaints (6) and how the parent copes with own symptoms may influence the health attitudes and behaviors of the child(7-10). This risk may be especially high if the parent suffers from health anxiety by proxy because the child is exposed to a particular preoccupation with and fear of illness and symptoms. For these reasons health anxiety by proxy is an important but neglected clinical phenomenon. Therefore, it is important to develop and test treatment targeting health anxiety by proxy.

Internet-based treatment is a relatively new approach that compares favourably with face-to-face treatment (15, 16). The Research Clinic for Functional Disorders and Psychosomatics (Research Clinic), Aarhus University Hospital (AUH) has recently developed an internet-based treatment program (iACT) for health anxiety based on principles from Acceptance and Commitment Therapy (ACT)(17). This treatment has shown promising results (14, 18) and is used as a template for the development of specialised treatment for parents with health anxiety by proxy. The treatment is called iACT-by proxy and is targeting parents' maladaptive anxiety-driven behaviour towards their child with focus on exposure therapy in the context of ACT principles.

The aim of the study is to test the feasibility and possible effect of the iACT- by proxy treatment program for health anxiety by proxy using a single-case experimental design.

Hypotheses

* Patients will report a significant decrease in selected self-report measures of health anxiety by proxy answered every other day when comparing the baseline period to the interven-tion period.
* Patient self-report measures of health anxiety by proxy, emotional distress, and illness perception and catastrophizing when the child has symptoms will have decreased after intervention.

Criteria for success of feasibility

* The treatment modules will be well received by the patients regarding format, length, content and contact to the therapist as measured by patient self-report on selected questions and with semi-structured interviews.
* Patients will log in to the modules on a weekly basis and will complete at least 6 out of 8 modules in the treatment. A module is complete when all text has been read in the module and corresponding exercises have been performed.
* Self-reported negative effects of participating are low.

Method

Participants and recruitment

The patients apply for participation in the project through the webpage www.helbredsangst.dk using NemID. On the webpage the patient will find information about health anxiety by proxy and the research project.

When logging in the participant is met with written information about participation and a following statement of consent giving permission to the health professionals in the project to directly collect health information from the patient record and use questionnaire data for research purposes in anonymised form. NemID is accepted as a digital signature by the Data Protection Agency. After the statement of consent, the participant is redirected to a questionnaire about physical and psychological symptoms, and personal background information. If the questionnaire is complete and the consent is signed the participant is self-referred. The participant will be invited to a video-assessment through e-boks.

Assessment

All participants are assessed using a shorter standardised diagnostic interview based on SCAN (Schedules for Clinical Assessment in Neuropsychiatry (21)) and supplemented with assessment of health anxiety by proxy using the HAPYS. The passed information from the patient record concerning the patients' somatic and psychiatric health information is necessary supplementary information for conducting a thorough assessment.

The interview is conducted using an encrypted link for a video-service hosted by the Central Denmark Region (rooms.rm.dk) which comply with the General Data Protection Regulation (GDPR). At the beginning of the interview, the health-professional ensures that the interview will be uninterrupted. The participant can have lay representative present during the interview if preferred.

Informed consent

All participants receive written and verbal information about the project. The participants receive the written information at self-referral. Verbal information is given by the health-professional performing the diagnostic assessment at the Research Clinic, AUH. They sign two consents; one when they complete the self-referral before the diagnostic interview, which gives the responsible investigators direct access to collect information from the electronic patient record for the purpose of using the participant's health information; and one consent when entering the research project after the diagnostic assessment.

Signing the final consent the participants enters the project, gives permission to publish the research data, and gives permission to being contacted during the study period. In order to uphold the treatment responsibility, the participant provides a phone number of a relative in case of suicide suspicion. The system allows the participant to log out and log in again at a later time providing the participant with the opportunity to reflect before signing the consent. If the consent is not signed within two weeks after the interview the participant will be excluded from the study.

Design

The single-case experimental study will be designed with multiple baselines comparing the individuals' baseline level of health anxiety by proxy with the level of health anxiety by proxy during and following participation in the treatment (19, 22). In a multiple baseline design, the participants have different baseline lengths but the same intervention and follow-up period. The baseline and intervention period serves as two study conditions, a control (baseline) and a treatment condition (intervention) with N equally spaced measurement occasions(19). The base-line length is randomly assigned to the participants and serves as each participants' own control-condition. This makes it possible to have a small number of participants. If the intervention shows effect a change in the anxiety level will be detected during the intervention period.

Measurements

All measures are self-report measures obtained through the secure web-based software platform for data collection REDCap (Research Electronic Data Capture)(23, 24) hosted at Aarhus University.

Assessment

* Short version of Schedules for Clinical Assessment in Neuropsychiatry (20, 21)
* The Health Anxiety by Proxy Scale (HAPYS) (Ingeman et al., submitted)

Primary outcome

The target measures of health anxiety by proxy are answered though a link in a SMS to the participants every other day from start of baseline to end of follow-up. The order of the items will be random each day. The target measures contain items of core characteristics of health anxiety by proxy which have been selected from the HAPYS based on the following:

Secondary outcome

Standardised self-report questionnaires will be answered four times during the study period (before baseline, right before treatment entry (end of baseline), end of treatment, and at 4-weeks follow-up.

Feasibility outcome

Participants are asked to provide feedback on format, length and content of the treatment program as well as on the contact to the therapist after each treatment-module and in a semi-structured phone-interview with the Ph.D.-student after treatment end.

Intervention

The treatment is an eight-week therapist-supported internet-based program based on written psychoeducation, audio-files, behavioural exposure exercises, homework and videos distributed in eight short modules.

Data analysis

Analysis will be divided into primary outcome and secondary outcome. The primary outcome will be analysed using visual analysis of plotting data and observing if the measures decreases at time of intervention entry (19). Further, using a Bayesian analysis of clinically significant change will quantify the evidence for the size and presence of an intervention effect (35, 36). The secondary outcome is analysed by determining Jacobsen's Reliable Change Index and from this determine that the change seen is not at result of measurement error and whether it is clinically significant(19, 37). The online free-text-answers and the interview on formalities and contact to therapist will be explored using thematic analysis focusing on all participant-experiences.

Funding

The Ph.D.-student and the Department of Child and Adolescent Psychiatry has initiated the research project in collaboration with the Research Clinic, AUH and received funding from numerous funds.

Ethics

The project is conducted in accordance to the rules in the Helsinki-Declaration. The project is registered under the Central Denmark Region's records of research projects (Den interne fortegnelse over forskningsprojekter ved Region Midt; 1-16-02-921-17).

There is no previous research data suggesting that internet-based treatment for health anxiety, anxiety or depression are associated with any form of risk (12, 14-16, 18).

Data protection

All information concerning the participants is protected by the data protection act and the data protection regulation. All personal data including name, telephone number and social security number is encrypted. The questionnaires are not personally identifiable, but have a random ID-number. The participants provide written informed consent to publish data in a single-case format where each participant's data is reported separately, but anonymized.

The platform hosting the treatment program was developed and programmed at the Research Clinic for Functional Disorders and Psychosomatics. All access to the server goes through an encrypted SSL-connection, and data pooling is being logged with IP and user-ID. NemID is used to log in to the platform. Access to the questionnaire data is only granted to researchers in the project and the data will be kept anonymously after project-end.

Project group

The project is conducted at the Research Clinic in collaboration with the Department of Child and Adolescent Psychiatry, AUH.

The project group consist of Katrine Ingeman Beck, psychologist (PhD student)1,2, Charlotte Ulrikka Rask, MD, professor, PhD1,2 (Main supervisor); Lisbeth Frostholm, head psychologist, associate professor, PhD3,2 (Co-supervisor); Kristi Wright, psychologist, associate professor, PhD4 (Co-supervisor); Ditte Hoffmann Jensen, psychologist, PhD3 (Co-supervisor).

1. Department of Child and Adolescent Psychiatry, AUH, Psychiatry, Aarhus, Denmark.
2. Department of Clinical Medicine, Aarhus University, Denmark
3. The Research Clinic, AUH, Aarhus, Denmark.
4. Department of Psychology, Faculty of Arts, University of Regina, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Parents of age
* Assessed with severe health anxiety by proxy
* At least one child under 18 years
* Healthy children without severe hospital-treatment-requiring diagnoses or disabilities
* Read, write and speak Danish

Exclusion Criteria:

* Comorbid diagnoses of substance abuse, bipolar disorder, psychotic disorders (ICD-10: F20-29) or autism spectrum disorder.
* Recently starting up psychotropic drug (with-in the last two months)
* Suicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
SMS-data | Up to 15 weeks
  Four questions assessing patients anxiety level is sent to the patient every day by sms.

SECONDARY OUTCOMES:
The health anxiety by proxy scale | Baseline, 1-3 weeks, 9-11 weeks, 13-15 weeks
  Self-report questionnaire assessing parent's worries about their child's health
The Adult Response to Children's Symptoms (ARCS) - parent form (revised) | Baseline, 1-3 weeks, 9-11 weeks, 13-15 weeks
  Self-report questionnaire assessing parent's reactions when their child has symptoms
Pain Catastrophizing Scale - parent version | Baseline, 1-3 weeks, 9-11 weeks, 13-15 weeks
  Self-report measure assessing parental catastrophic thinking when their child is in pain.
The Whiteley-6 Index | Baseline, 1-3 weeks, 9-11 weeks, 13-15 weeks
  Self-report measure assessing health related worries
SCL-8 (emotional distress) | Baseline, 1-3 weeks, 9-11 weeks, 13-15 weeks
  Self-report measure assessing emotional distress
WHO-5 Well-Being Index | Baseline, 1-3 weeks, 9-11 weeks, 13-15 weeks
  Self-report measure assessing general well-being
Experience of Service Questionnaire | 13-15 weeks
  Self-report measure assessing the experience of the treatment received
The Negative Effects Questionnaire | 13-15 weeks
  Self-report measure assessing negative effects of psychotherapy
Internet Evaluation and Utility Questionnaire | 13-15 weeks
  Self-report measure assessing the dilivery of internet-based treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ulrikka Rask, Med.Dr, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University hospital, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article will be available after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. The type of analyses are defined by the aims in the approved proposal.
  Proposals may be submitted up to 36 months following article publication. Proposals should be directed to katbec@rm.dk. To gain access, data requestors will need to sign a data access agreement. After 36 months the data will be available in a data warehouse but without investigator support.

REFERENCES:
- [Background] Lockhart E. Health anxiety in children and parents. BMJ. 2016 May 24;353:i2891. doi: 10.1136/bmj.i2891. No abstract available. PMID 27222022
- [Background] Thorgaard MV, Frostholm L, Walker L, Jensen JS, Morina B, Lindegaard H, Salomonsen L, Rask CU. Health anxiety by proxy in women with severe health anxiety: A case control study. J Anxiety Disord. 2017 Dec;52:8-14. doi: 10.1016/j.janxdis.2017.09.001. Epub 2017 Sep 11. PMID 28950218
- [Background] Thorgaard MV, Frostholm L, Rask CU. Childhood and family factors in the development of health anxiety: A systematic review. Children's Health Care. 2017:1-41
- [Background] Thorgaard MV, Frostholm L, Walker LS, Stengaard-Pedersen K, Karlsson MM, Jensen JS, Fink P, Rask CU. Effects of maternal health anxiety on children's health complaints, emotional symptoms, and quality of life. Eur Child Adolesc Psychiatry. 2017 May;26(5):591-601. doi: 10.1007/s00787-016-0927-1. Epub 2016 Dec 1. PMID 27909834
- [Background] Walker LS, Williams SE, Smith CA, Garber J, Van Slyke DA, Lipani TA. Parent attention versus distraction: impact on symptom complaints by children with and without chronic functional abdominal pain. Pain. 2006 May;122(1-2):43-52. doi: 10.1016/j.pain.2005.12.020. Epub 2006 Feb 21. PMID 16495006
- [Background] Jamison RN, Walker LS. Illness behavior in children of chronic pain patients. Int J Psychiatry Med. 1992;22(4):329-42. doi: 10.2190/AMAN-GJ29-4N1C-6JR2. PMID 1293062
- [Background] Craig TK, Cox AD, Klein K. Intergenerational transmission of somatization behaviour: a study of chronic somatizers and their children. Psychol Med. 2002 Jul;32(5):805-16. doi: 10.1017/s0033291702005846. PMID 12171375
- [Background] Wright KD, Reiser SJ, Delparte CA. The relationship between childhood health anxiety, parent health anxiety, and associated constructs. J Health Psychol. 2017 Apr;22(5):617-626. doi: 10.1177/1359105315610669. Epub 2015 Oct 14. PMID 26466851
- [Background] Koteles F, Freyler A, Kokonyei G, Bardos G. Family background of modern health worries, somatosensory amplification, and health anxiety: A questionnaire study. J Health Psychol. 2015 Dec;20(12):1549-57. doi: 10.1177/1359105313516661. Epub 2014 Jan 8. PMID 24406331
- [Background] Hedman E, Andersson G, Andersson E, Ljotsson B, Ruck C, Asmundson GJ, Lindefors N. Internet-based cognitive-behavioural therapy for severe health anxiety: randomised controlled trial. Br J Psychiatry. 2011 Mar;198(3):230-6. doi: 10.1192/bjp.bp.110.086843. PMID 21357882
- [Background] Hoffmann D, Rask CU, Hedman-Lagerlöf E, Jensen JS, Frostholm L. Internet-delivered psychological treatment for patients with health anxiety: Results from a randomized, controlled trial. Journal of psychosomatic research. 2019;121:113-.
- [Background] Andersson G. Using the Internet to provide cognitive behaviour therapy. Behav Res Ther. 2009 Mar;47(3):175-80. doi: 10.1016/j.brat.2009.01.010. Epub 2009 Feb 20. PMID 19230862
- [Background] Cuijpers P, Marks IM, van Straten A, Cavanagh K, Gega L, Andersson G. Computer-aided psychotherapy for anxiety disorders: a meta-analytic review. Cogn Behav Ther. 2009;38(2):66-82. doi: 10.1080/16506070802694776. PMID 20183688
- [Background] Hayes SC, Strosahl K, Wilson KG. Acceptance and commitment therapy : the process and practice of mindful change. 2. ed. ed. New York: Guilford Press; 2012. 402
- [Background] Hoffmann D, Rask CU, Hedman-Lagerlof E, Jensen JS, Frostholm L. Efficacy of internet-delivered acceptance and commitment therapy for severe health anxiety: results from a randomized, controlled trial. Psychol Med. 2021 Nov;51(15):2685-2695. doi: 10.1017/S0033291720001312. Epub 2020 May 14. PMID 32404226
- [Background] Morley S. Single-Case Methods in Clinical Psychology: A Practical Guide. 1 ed. Milton: Routledge; 2018.
- [Background] Hoffmann D, Rask CU, Hedman-Lagerlof E, Eilenberg T, Frostholm L. Accuracy of self-referral in health anxiety: comparison of patients self-referring to internet-delivered treatment versus patients clinician-referred to face-to-face treatment. BJPsych Open. 2019 Sep 9;5(5):e80. doi: 10.1192/bjo.2019.54. PMID 31496462
- [Background] Schedules for clinical assessment in neuropsychiatry : Manual. Version 2 ed. Geneva: WHO; 1994. 331 p.
- [Background] Tate RL, Perdices M, Rosenkoetter U, Shadish W, Vohra S, Barlow DH, Horner R, Kazdin A, Kratochwill T, McDonald S, Sampson M, Shamseer L, Togher L, Albin R, Backman C, Douglas J, Evans JJ, Gast D, Manolov R, Mitchell G, Nickels L, Nikles J, Ownsworth T, Rose M, Schmid CH, Wilson B. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) 2016 Statement. Am J Occup Ther. 2016 Jul-Aug;70(4):7004320010p1-11. doi: 10.5014/ajot.2016.704002. PMID 27294998
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] de Vries RM, Hartogs BM, Morey RD. A Tutorial on Computing Bayes Factors for Single-Subject Designs. Behav Ther. 2015 Nov;46(6):809-23. doi: 10.1016/j.beth.2014.09.013. Epub 2014 Oct 7. PMID 26520223
- [Background] de Vries RM, Meijer RR, van Bruggen V, Morey RD. Improving the analysis of routine outcome measurement data: what a Bayesian approach can do for you. Int J Methods Psychiatr Res. 2016 Sep;25(3):155-67. doi: 10.1002/mpr.1496. Epub 2015 Oct 8. PMID 26449152
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Derived] Ingeman K, Frostholm L, Wellnitz KB, Wright K, Frydendal DH, Onghena P, Rask CU. Internet-Delivered Therapy for Parents With Health Anxiety by Proxy: Protocol for a Single-Case Experimental Design Study. JMIR Res Protoc. 2023 Nov 24;12:e46927. doi: 10.2196/46927. PMID 37999936

DOCUMENTS (1):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT04830605/Prot_000.pdf